CLINICAL TRIAL: NCT01580787
Title: Functional Improvement in Patients With Parkinson's Disease After Training in Real or Virtual Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sao Camilo University Center (Other)
Responsible Party: Principal Investigator, Jose Eduardo Pompeu, Clinical Professor, Sao Camilo University Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: saocamilo-sp
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Parkinson´s Disease
Keywords: Parkinson´s disease; Postural Balance; virtual reality
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual Reality Training (Experimental): The virtual reality training was done by experimental group with ten games of Nintendo Wii Fit.
  Interventions: Device: Balance Training with Nintendo Wii Fit
- Physical Therapy (Active Comparator): The Control Group was trained by conventional Physical Therapy exercises.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Device: Balance Training with Nintendo Wii Fit — The participants of the study trained 10 balance games during 14 sessions.
  Arms: Virtual Reality Training
Other: Physical Therapy — Patients of the control group was trained with balance exercises.
  Arms: Physical Therapy

SUMMARY:
The objective of this work was to compare the effects of two balance training programs, one Nintendo Wii Fit-based and the other traditionally-based without the use of a gaming system, on the balance, functionality and cognition of patients with Parkinson´s disease. It was a prospective, single blinded, randomized clinical trial performed at Brazil Parkinson Association and Center of Research of the courses of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University. 32 patients with Parkinson´s disease on stages 1 and 2,5 of Hoehn e Yahr participated of this work. Patients were randomized in control and experimental group, 16 each one.

The study was finished at december 2011.

DETAILED DESCRIPTION:
The objective of this work was to compare the effects of two balance training programs, one Nintendo Wii Fit-based and the other traditionally-based without the use of a gaming system, on the balance, functionality and cognition of patients with Parkinson´s disease. It was a prospective, single blinded, randomized clinical trial performed at Brazil Parkinson Association and Center of Research of the courses of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University. 32 patients with Parkinson´s disease on stages 1 and 2,5 of Hoehn e Yahr participated of this work. Patients were randomized in control and experimental group, 16 each one. Both groups performed 14 training sessions, twice a week, for seven weeks. Each session was composed of a 30 minute-global-exercise series including stretching, muscle strengthen and axial mobility exercises. After this, both groups performed more 30 minutes of balance training: the control group performed balance exercises without external cues, visual or auditory feedbacks or cognitive stimulations; the experimental group performed the balance training with 10 Wii Fit games which stimulated motor and cognitive functions. The main outcome measures were: (1) Unified Parkinson´s Disease Rating Scale (UPDRS); (2) Berg Balance Scale (BBS); (3) Unipedal Stance Test (UST) and (4) Montreal Cognitive Assessment (MoCA). The statistical analysis was done by repeated measures ANOVA in order to assess the possible differences among the analyzed variables. Both groups showed improvement in the section II of UPDRS, BBS, UST and MoCA. Patients with Parkinson´s disease showed balance and cognitive improvement with positive repercussion on daily living activities after 14 sessions of balance training without additional advantages to the virtual training.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson´s disease
* both gender
* on stages 1 and 2,5 of Hoehn e Yahr

Exclusion Criteria:

* depression
* cognitive impairment
* deficits of visual acuity
* Score on Berg Balance Scale under 46

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
UNIFIED PARKINSON'S DISEASE RATING SCALE | 08/2011 (up to 2 years)
  The scale assesses the functional status of patients with parksinon´s disease, including the independency of daily activities, mood, secondary effects of medications and motor complications.

SECONDARY OUTCOMES:
Berg Balance Scale | 08/2011 (up to 2 years)
  Berg Balance Scale assesses the functional balance of patients with Parkinson´s disease. It is a clinic assessment of patient that evaluates the performance of patient to stand up and sit down, turn on and step, among others situations.

CONTACTS AND LOCATIONS:
Overall Officials: José E Pompeu, PhD, Principal Investigator — Sao Camilo University Center

REFERENCES:
- [Derived] Pompeu JE, Mendes FA, Silva KG, Lobo AM, Oliveira Tde P, Zomignani AP, Piemonte ME. Effect of Nintendo Wii-based motor and cognitive training on activities of daily living in patients with Parkinson's disease: a randomised clinical trial. Physiotherapy. 2012 Sep;98(3):196-204. doi: 10.1016/j.physio.2012.06.004. Epub 2012 Jul 25. PMID 22898575